CLINICAL TRIAL: NCT05298033
Title: Study of Efficacy, Safety and Tolerability of Crisaborole and PF-07038124 With and Without NBUVB in Vitiligo: A Phase 2A Randomized, Double-Blind, Vehicle-Controlled Clinical Trial
Brief Title: Study of Efficacy, Safety and Tolerability of Crisaborole and PF-07038124 With and Without NBUVB in Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-4837
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Vitiligo
Keywords: Vitiligo; PDE-4 inhibitor; Phototherapy; Repigmentation
MeSH Terms: conditions — Vitiligo | interventions — crisaborole; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (6):
- Active NBUVB plus Crisaborole 2% topical ointment (Experimental): 12 participants will receive 6 months of treatment with crisaborole 2% topical along with 6 months of treatment with active NBUVB
  Interventions: Drug: Crisaborole 2 % Topical Ointment; Device: NBUVB phototherapy
- Active NBUVB plus PF-07038124 0.01% topical ointment (Experimental): 12 participants will receive 6 months of treatment with active NBUVB, to be combined with 3 months of treatment with PF-07038124 0.01% topical ointment followed by 3 months of vehicle ointment
  Interventions: Drug: PF-07038124 0.01% topical ointment; Device: NBUVB phototherapy; Drug: Vehicle
- Active NBUVB plus vehicle ointment (Active Comparator): 8 participants will receive 6 months of treatment with active NBUVB combined with 6 months of vehicle ointment application
  Interventions: Device: NBUVB phototherapy; Drug: Vehicle
- Sham phototherapy plus crisaborole 2% topical ointment (Experimental): 12 participants will receive 6 months of treatment with crisaborole 2% topical ointment combined with 6 months of sham phototherapy
  Interventions: Drug: Crisaborole 2 % Topical Ointment; Device: Sham phototherapy
- Sham phototherapy plus PF-07038124 0.01% topical ointment (Experimental): 12 participants will receive 3 months of treatment with PF-07038124 0.01% topical ointment, followed by 3 months of vehicle ointment, along with 6 months of sham phototherapy
  Interventions: Drug: PF-07038124 0.01% topical ointment; Device: Sham phototherapy; Drug: Vehicle
- Sham phototherapy plus vehicle ointment (Placebo Comparator): 8 participants will receive 6 months of sham phototherapy combined with 6 months of vehicle ointment application
  Interventions: Device: Sham phototherapy; Drug: Vehicle

INTERVENTIONS:
Drug: Crisaborole 2 % Topical Ointment — Twice daily crisaborole 2% topical ointment
  Other Names: Eucrisa
  Arms: Active NBUVB plus Crisaborole 2% topical ointment; Sham phototherapy plus crisaborole 2% topical ointment
Drug: PF-07038124 0.01% topical ointment — Twice daily PF-07038124 0.01% topical ointment
  Arms: Active NBUVB plus PF-07038124 0.01% topical ointment; Sham phototherapy plus PF-07038124 0.01% topical ointment
Device: NBUVB phototherapy — Home narrow band UVB phototherapy exposure sessions 3 times per week
  Other Names: Narrow band UVB
  Arms: Active NBUVB plus Crisaborole 2% topical ointment; Active NBUVB plus PF-07038124 0.01% topical ointment; Active NBUVB plus vehicle ointment
Device: Sham phototherapy — Non-NBUVB visible light radiation exposure sessions 3 times per week
  Arms: Sham phototherapy plus PF-07038124 0.01% topical ointment; Sham phototherapy plus crisaborole 2% topical ointment; Sham phototherapy plus vehicle ointment
Drug: Vehicle — Twice daily vehicle ointment
  Arms: Active NBUVB plus PF-07038124 0.01% topical ointment; Active NBUVB plus vehicle ointment; Sham phototherapy plus PF-07038124 0.01% topical ointment; Sham phototherapy plus vehicle ointment

SUMMARY:
This is a phase 2A clinical trial designed to test the pro-melanogenic and anti-inflammatory role of phosphodiesterase-4 inhibitors (PDE4i), alone and in combination with active narrow band UVB (NBUVB), in vitiligo lesions. This is a double-blind, randomized controlled trial (RCT) with six study arms. The goal is for 64 participants to be recruited and complete the study.

ELIGIBILITY:
Inclusion Criteria:

Active or stable non-segmental vitiligo at Screening and Baseline visits:

* A clinical diagnosis of non-segmental vitiligo (vitiligo vulgaris or acrofacial vitiligo) for at least 3 months, AND
* Body Surface Area affected (BSA) involvement 3%-90%, excluding involvement of scalp, palms of the hands, soles of the feet, AND
* BSA >= 0.25% involvement of the facial area, AND
* Minimum Facial Vitiligo Area Scoring Index (F-VASI) >=0.25% and Total VASI >=3%
* Must agree that the treatment area will involve 3%-25% BSA
* If receiving concomitant medication for any reason other than vitiligo, must be on a stable regimen (no new drug or dosage changes within 7 days of baseline visit) and willing to remain on stable regimen for duration of the study
* Must agree to stop all other treatments for vitiligo from screening through 1 week after discontinuation of study drug treatment
* Must be capable of giving signed informed consent and comply with the requirements and restrictions as listed in the informed consent document and protocol
* Must agree to avoid exposure to the sun as much as possible and not to use tanning booths, sun lamps, or other ultraviolet light sources other than requested by the study team during the study

Exclusion Criteria:

* Pregnant or breastfeeding females
* Females of childbearing potential who are unwilling or unable to use contraception for the duration of the study and for at least 28 days after the last dose of study intervention
* Other types of vitiligo that do not meet criteria for active or stable or non-segmental vitiligo, including segmental, mucosal, focal, and mixed vitiligo, and those with vitiligo universalis
* Active forms of other hypo- or depigmentation, as detailed in the protocol
* Active forms of inflammatory skin disease(s) associated with hypo- or depigmentation at the time of screening or baseline that, in the opinion of the investigator, would interfere with evaluation of vitiligo or response to treatment
* Leukotrichia in more than 33% of the facial area affected with vitiligo lesions OR leukotrichia in more than 33% of the total BSA affected with vitiligo lesions
* History of transplantation procedure for vitiligo at any point
* History of any skin bleaching treatment for vitiligo or other dermatoses at any point
* Active acute or chronic skin infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to first drug application (baseline), OR superficial skin infections within 2 weeks prior to first drug application (NOTE: MAY BE RESCREENED AFTER INFECTION RESOLUTION)
* Known history of severe allergic or anaphylactoid reaction to any PDE4 inhibitors or lidocaine
* Documented lack of response to prior PDE4 inhibitor therapy
* Presence of other severe, progressive, or uncontrolled diseases, including but not limited to renal, hepatic, cardiac, pulmonary, endocrine, immunological/rheumatological, hematological, gastrointestinal, metabolic, neurologic, psychiatric, immunodeficiency (including HIV positive serology), OR significant laboratory abnormalities that would increase risk associated with study participation or interfere with interpretation of study results, or in the opinion of the investigator, the participant is inappropriate for entry into the study, or unwilling/unable to comply with protocol-specified assessments and lifestyle considerations
* Any malignancies or history of skin malignancies, excluding adequately treated or excised non-metastatic basal cell or squamous cell skin cancer, or cervical carcinoma in situ
* Significant trauma or major surgery 1 month prior to screening or considered in imminent need of surgery during the study
* Alcohol or substance abuse within 6 months of screening that in the opinion of the investigator would preclude participation or adherence in the study
* Previous administration of an investigational drug or vaccine occurring within 30 days preceding the first application of study drug used in this study
* Any biologic or immune-modulating agent (including oral JAK inhibitors, PDE4i, other immunosuppressive agents such as oral corticosteroids, calcineurin inhibitors, azathioprine, mycophenolate mofetil) requires a washout period of 8 weeks before screening and through the final safety follow-up visit
* Any topical treatment (such as topical steroids, calcineurin inhibitors, vitamin D analogs, JAK inhibitors, PDE4i) requires a washout period of 2 weeks before screening visit and through the final safety follow-up visit
* Ultraviolet light exposure, including UVB/UVA/PUVA delivered by booth/excimer laser, or tanning bed exposure, requires a washout period of 8 weeks before screening and through the final safety follow-up visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving at 50% or greater improvement from baseline in facial Vitiligo Area Scoring Index (F)-VASI | 6 months (week 24)
  Assessment of facial repigmentation via changes in depigmented areas

SECONDARY OUTCOMES:
Proportion of participants achieving 90% or greater improvement from baseline in F-VASI | 6 months (week 24)
Proportion of participants achieving 50% or greater improvement from baseline in total (T)-VASI | 6 months (week 24)
Proportion of participants achieving a Vitiligo Noticeability Scale (VNS) rating of "a lot less noticeable" or "no longer noticeable" | 6 months (week 24)
Percentage change from baseline in facial segment of Body Surface Area affected (F-BSA) | 6 months (24 weeks)

OTHER OUTCOMES:
Quantification of pigment via Fontana-Masson staining | Baseline (day 0, pre-treatment) and 3 months (12 weeks)
  Molecular outcome: using skin biopsies treated with PDE4i with/without active NBUVB
Assessment of melanocyte population expansion via immunohistochemistry (IHC) studies | Baseline (day 0, pre-treatment) and 3 months (12 weeks)
  Molecular outcome: using skin biopsies treated with PDE4i with/without active NBUVB
Assessment of percent change from baseline in serum key inflammatory chemokines | Baseline (pre-treatment) and at 3 months (12 weeks) and 6 months (24 weeks)
  Molecular outcome: using samples for serum measurements of IFN-gamma, IL-15, CXCL-9, CXCL-10, which have been implicated in vitiligo pathogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Stanca Birlea, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz - Clinical and Translational Research Centers, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No